CLINICAL TRIAL: NCT04675697
Title: Anlotinib Plus Platinum-etoposide in First-line Treatment of Extensive-stage Small-cell Lung Cancer: a Single-arm Phase II Trial
Brief Title: Anlotinib Plus Platinum-etoposide in First-line of Extensive-stage Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019010023
Record Dates: First submitted 2020-12-02; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib+EP (Experimental)
  Interventions: Drug: Platinum-etoposide+Anlotinib

INTERVENTIONS:
Drug: Platinum-etoposide+Anlotinib — Platinum-etoposide regiment consisted of etoposide 100mg/m2, d1~3 of 21-day cycle, with investigators' choice of either cisplatin (75-80mg/m2, Q3W) or carboplatin (AUC=5~6, Q3W). Anlotinib treated of 12mg Qd from day 1 to 14 of a 21-day cycle. Eligible patients received anlotinib plus platinum-etoposide for 4~6 cycles, and followed by maintenance therapy with Anlotinib. The efficacy was evaluated every 6 weeks (2 cycles) through treatment.

SUMMARY:
Anlotinib is a novel multi-target tyrosine kinase inhibitor (TKI) for tumor angiogenesis and tumor cell proliferation. The efficacy of Anlotinib as a third-line or beyond therapy for SCLC was confirmed in the ALTER1202 trial. The aim of this trial was to investigate the prognostic value of Anlotinib plus platinum-etoposide in first-line treatment of extensive-stage SCLC patients.

DETAILED DESCRIPTION:
This single-arm phase II trial enrolled extensive-stage SCLC patients without prior systematic chemotherapy or immunity checkpoint inhibitors therapy at Xiangya hospital, Central South University from Aug 15, 2018 to Oct 7, 2020.The study was done in accordance with the International Conference on Harmonisation good clinical practice guidelines, the Declaration of Helsinki, and applicable local regulations with approval from an independent ethics committee or institutional review boards.

Eligible patients were age 18-70 years with histologically confirmed extensive-stage small-cell lung cancer as defined according to the staging standard introduced by the Veterans Administration Lung Study Group (VALG), measurable according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1), and an Eastern Cooperative Oncology Group (ECOG) performance-status (PS) score of 0 or 1, who had not received previous systemic treatment for extensive-stage small-cell lung cancer and were expected survival time ≥3 months. Patients with treated asymptomatic central nervous system (CNS) metastases were eligible under some circumstance (see the Supplementary Appendix). Key exclusion criteria were a history of mixed small cell carcinoma and non-small cell carcinoma and with active central nervous system (CNS) metastasis and/or cancerous meningitis during screenings.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged 18 to 70 years old;
* Rated as grade 0 to 2 in ECOG whole-body status (PS), or grade 3 to 4 if induced by SCLC;
* Of the expected survival no less than 3 months;
* With extensive-stage SLCL diagnosed pathologically (according to the VALG staging standard introduced by the Veterans Administration Lung Study Group), and having a measurable lesion (a tumor lesion of ≥ 10mm in long diameter in CT scanning, or a lymph node lesion of ≥ 15mm in short diameter in CT scanning, which had not received radiotherapy, cryotherapy or other local therapies, according to the RECIST1.1 standard);
* Having not received chemotherapy or immunotherapy;
* Some patients who have received radiotherapy can be included as long as the radiotherapy area in them is smaller than 25% of the bone marrow area, they haven't undergone total pelvic or chest radiation, their previous radiotherapy ended at least 4 weeks before the inclusion, they have recovered from radiotherapy-induced acute toxicity reaction, and the local lesion that underwent radiotherapy in them is not included in the measurable lesion, unless significant progress was observed in the lesion after the last radiotherapy.
* Patients included should also have normal major organ functions, that is, their organs should meet the following criteria:

  1. Blood routine examination criteria: ANC ≥ 1.5 × 109/L, PLT ≥ 100 × 109/L and Hb≥100g/L (no blood transfusion or blood products in 14 days, and no G-CSF or other hematopoietic stimulant corrections).
  2. Biochemical examination criteria: TBIL < 1.5 × ULN, ALT, AST and ALP < 2.5 × ULN, BUN and Cr ≤ 1 × ULN, or endogenous creatinine clearance rate ≥ 50ml/min.
* Females of childbearing age should have taken reliable contraceptives or have had a negative pregnancy test (serum or urine) result 7 days before inclusion, and should be willing to take appropriate contraception measures during the study and in 8 weeks after the last administration of the treatment drug. Males should agree to take appropriate contraception measures during the study and in 8 weeks after the last administration of the treatment drug or have undergone sterilization operation.
* Subjects should voluntarily participate in the study, sign the Informed Consent, and be well compliant and cooperative in follow-up visits.

Exclusion Criteria:

* Having mixed small cell carcinoma and non-small cell carcinoma;
* Having active central nervous system (CNS) metastases and/or cancerous meningitis or found to have active central nervous system (CNS) metastases and/or cancerous meningitis in examinations during the screening stage. Patients can be included in the study as long as they: (1) Have asymptomatic brain metastases (without progressive central nervous system symptoms induced by brain metastases, requiring no corticosteroids, and having the lesion size ≤ 1.5cm), provided that they should undergo regular brain imaging examinations for the diseased site; (2) Have been treated and are in stable status, have no imaging evidence for new or enlarged brain metastases at least 2 weeks after brain metastasis treatment, and have discontinued steroids or anticonvulsants at least 14 days before the therapy of the study starts.
* Patients whose imaging findings showed invaded central great vessels or obvious pulmonary cavity or necrotizing tumor should be excluded.
* Patients with hypertension who are taking two or more antihypertensive drugs should be excluded.
* Patients having the following should be excluded: Cardiovascular diseases: Myocardial ischemia or myocardial infarction or grade II or above, uncontrolled arrhythmias, new functions of grade III to IV, or cardiac ejection fraction < 50%;
* Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds, or APTT > 1.5ULN), prone to bleeding or receiving thrombolytic or anticoagulant therapy;
* Had significant cough blood or daily hemoptysis of 2.5ml or more in 2 months before the inclusion;
* Having bleeding symptoms or definite bleeding tendency of significant clinical significance, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ or above at baseline, or vasculitis, in 3 months before the inclusion;
* Having developed artery/venous thrombosis in 12 months before the inclusion;
* With known hereditary or acquired bleeding and thrombosis tendency;
* Having a wound or fracture that has cannot be healed for a long time;
* Having received major surgery or had severe traumatic injury, fracture or ulcer in 4 weeks before the inclusion;
* Subject to factors that significantly affect the absorption of oral medication;
* Having developed abdominal fistula, gastrointestinal perforation or abdominal abscess in 6 months before the inclusion;
* Having the urine routine result suggest urine protein ≥++, or confirmed the 24-hour urine protein amount ≥ 1.0g;
* With serous membrane effusion that is with clinical symptoms and requires symptomatic treatment;
* With active infections that require antimicrobial treatment;
* Having a history of psychotropic drug abuse and unable to quit or with a mental disorder;
* Having participated in other clinical trials on anti-tumor drugs 4 weeks before the inclusion;
* Previously or currently having other incurable malignancies;
* Having received over-potent CYP3A4 inhibitor treatment in 7 days before the inclusion, or have received over-potent CYP3A4 inducer treatment in 12 days before the inclusion.
* Pregnant or lactating women who are fertile but are unwilling or unable to take effective contraception measures should be excluded.
* Patients as determined by researchers to be subject to other conditions that may clinically affect the conduct or outcome of the study should be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 1 year
  progression-free survival
ORR | up to 1 year
  objective response rate (ORR, CR+PR)

SECONDARY OUTCOMES:
OS | From randomization until death (up to 15 months)
  overall survival
DCR | At the end of every 2 cycles (each cycle is 21 days)，through treatment，up to 1 year
  disease control rate (DCR, CR+PR+SD)
DoR | At the end of every 2 cycles (each cycle is 21 days)，through treatment，up to 1 year
  duration of remission

CONTACTS AND LOCATIONS:
Overall Officials: Huaping S Yang, M.D, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Deng P, Hu C, Chen C, Cao L, Gu Q, An J, Qin L, Li M, He B, Jiang J, Yang H. Anlotinib plus platinum-etoposide as a first-line treatment for extensive-stage small cell lung cancer: A single-arm trial. Cancer Med. 2022 Oct;11(19):3563-3571. doi: 10.1002/cam4.4736. Epub 2022 May 8. PMID 35526266